CLINICAL TRIAL: NCT00237068
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Gastroesophageal Reflux Disease Therapy ( Lansoprazole; Solutab) in the Management of Childhood Asthma
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Study of Gastroesophageal Reflux Disease Therapy.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Emory University (Other)
Responsible Party: Benjamin Gold, MD, Emory University
Organization: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: GERD AsthmaStudy
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Asthma
Keywords: Gastroesophageal Reflux
MeSH Terms: conditions — Asthma; Gastroesophageal Reflux | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lansoprazole; Solutab — 15 and 30 mg doses of dissolvable tablet, 2 tablets daily for one year
  Other Names: Prevacid

SUMMARY:
Asthma and gastroesophageal reflux disease (GERD) are common disorders, which although are not usually lethal, both have high morbidity, and high healthcare costs. Recent studies have demonstrated that asthma and GERD often co-exists, and that this co-existence is more frequent than just chance. Therefore, studies that characterize associations between these conditions, and, help in the development of interventions will positively impact the outcomes of these patients, which are critically needed.

Subjects that participate in this study are required to be between the ages of 4-11 years old. This protocol proposes to enroll 100 children with asthma, on inhaled steroids who have poor asthma control, defined on the basis of frequent symptoms, excessive beta-agonists use, or frequent asthma episodes.

The purpose of this research study is to:

1. Determine, whether children with symptomatic, poorly controlled, asthma assigned to treatment with a PPI( Proton Pump Inhibitor), have fewer asthma exacerbations than similar participants assigned to placebo for a similar duration of time
2. Determine whether children treated with Lansoprazole ( i.e., proton pump inhibitor): have a longer time to first exacerbation, have improved lung function, improved asthma symptom scores, improved quality of life, decreased rescue inhaler use, or other asthma medications, reduced emergency room/urgent care/ physician office visits that are asthma related.
3. Determine whether a subgroup of symptomatic asthmatics, who show a greater benefit from PPI's, can be identified.

DETAILED DESCRIPTION:
GERD and asthma likely co-exist, and may be pathogenetically linked. However, it is controversial whether GERD per se is an important risk factor for severe asthma, and whether treatment of GERD and/or GERD symptoms improves asthma control. In addition, there are no published data on how often asthmatics are treated with the anti-secretory agents proton pump inhibitors (PPIs) for GERD. However, a preliminary survey from the American Lung Association's Asthma Clinical Research Centers consortium show diverse practice patterns among clinics with about 15% of children and 20% - 30% of adults being prescribed medical treatment (unpublished data).

The NIH Expert Panel on The Diagnosis and Management of Asthma, recommends that "…for patients with poorly controlled asthma, particularly with a nocturnal component, investigation for gastroesophageal reflux may be warranted even in the absence of suggestive symptoms". The American Thoracic Society (ATS) workshop on severe refractory asthma, concluded that GERD "…could contribute to the severity" of asthma and recommended that all patients with severe refractory asthma undergo esophageal pH probe monitoring to evaluate for the presence of GERD". Noticeably absent in both of these "expert panel" documents were randomized placebo controlled trial data in all populations, and properly designed clinical trial information in the pediatric population with clear case and control definitions of GERD and asthma. The American Gastroenterological Association recommends ambulatory pH probe monitoring in adult patients with reflux-triggered asthma; but, to date has developed no recommendations for children 20. While these are reasonable recommendations, there is no convincing evidence that GERD is more common in patients with severe asthma than mild asthma, or that treatment of reflux can decrease asthma severity. PPIs, the most effective treatment for GERD (i.e., resolve both symptoms and mucosal disease), have a retail cost between $100 and $153 per month. However, recent hospital data demonstrates that anti-reflux surgery is being performed at an increasing rate in children with respiratory manifestations of their GERD at a sizeable cost and with no long term outcome studies to date. Thus, it can be estimated that the cost for diagnosing and treating GERD in symptomatic asthmatics ranges from $1 to $8 billion dollars per year if all poorly controlled asthmatics were both investigated and treated. Therefore, randomized controlled clinical trials are critically needed to reduce overall healthcare costs and the public health burden of these two chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

4-11 years Informed Consent/ Assent Asthma Clinically normal laboratory results and physical exam

Exclusion Criteria:

Unable or unwilling to give informed consent Unable to comply with study protocol Any preexisting condition that would require A PPI for a period of 6 months or more and/other major chronic illnesses.

Drug Allergies toPPI. At High risk for non-compliance and/or adherence.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
One of the aims of this trial is to see if we can demonstrate a significant response to acid-suppression therapy in a group of poorly controlled childhood asthmatics using the number of asthma exacerbations as outcome variables. | 3 year

SECONDARY OUTCOMES:
A major unanswered question is whether severity or frequency of asthma is related to the response to anti-reflux treatment. | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D. Gold, MD., Principal Investigator — Emory University School of Medicine / Pediatrics
Locations (3):
- United States (3):
  - Emory Children's Center, Atlanta, Georgia
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Georgia Pediatric Pulmonology Associates/ CHOA, Atlanta, Georgia